CLINICAL TRIAL: NCT06601387
Title: Evaluation of Choledochoduodonostomy Vs Hepaticojejunostomy in Patients with Choledocholithiasis Indicated for Shunt .
Brief Title: Evaluation of Choledochoduodonostomy Vs Hepaticojejunostomy in Paients with Choledocholithiasis Indicated for Shunt.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamed Ahmed Hassan Aly (Other)
Responsible Party: Sponsor-Investigator, Mohamed Ahmed Hassan Aly, Assistant lecturer general surgery department, Assiut University
Organization: Assiut University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Surgery for common bile duct
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-09

CONDITIONS: Recurrent Common Bile Duct Stones
Keywords: Choledochoduodonostomy; Hepaticojejunostomy; Choledocholithiasis
MeSH Terms: conditions — Choledocholithiasis

STUDY DESIGN:
Intervention Model Description: comparative prospective study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group 1 of patients (Other): recurrent CBD Stones.
  Interventions: Procedure: choledochoduodonostomy
- group 2 of patients (Other): recurrent CBD stones
  Interventions: Procedure: hepaticojejunostomy

INTERVENTIONS:
Procedure: choledochoduodonostomy — surgical drainage procedures
  Arms: group 1 of patients
Procedure: hepaticojejunostomy — surgical intervention
  Arms: group 2 of patients

SUMMARY:
A biliary-enteric anastomosis can be needed for a number of indications, including malignant or pre-malignant biliary diseases, benign biliary stenosis, bile duct injury, and complex choledocholithiasis. Choledochoduodenostomy is the most simple form of biliary-digestive anastomosis, with only minimal alteration to the normal anatomy. Due to the reported specific complications of choledochoduodenostomy, such as sump syndrome and gastritis caused by biliary reflux, creation of a HJ was preferred in the past decades . A Roux-en-Y hepaticojejunostomy (HJ) does not cause sump syndrome and only rarely reflux gastritis, but the procedure is more extensive, requiring an additional jejuno-jejunostomy .Especially for patients with extensive intra-abdominal adhesions or with a history of small bowel resections, the creation of a Roux-en-Y limb might pose a problem. Some recent publications have concluded that CD leads to acceptable surgical outcome, with low reported incidences of sump syndrome and reflux gastritis. However, these studies do not make a direct comparison between CD and HJ. Especially comparisons of long-term outcomes between CD and HJ are lacking.

DETAILED DESCRIPTION:
There are 2 options are available: Choledochoduodonostomy or Roux-en-Y choledochojejunostomy. Both can be accomplished via a laparoscopic approach; however, thereis no consensus to which is best due to a paucity of data comparing the techniques.

Choice of operation is largely left up to the individual surgeon. Athough performed infrequently for benign biliary disease, biliary bypass operations are fundamental for any surgeon and are considered a core operation by the American College of Surgeons for any general surgery resident. In our study we are going to describe in detail our technique and outcomes when used for choledocholethiasis.

ELIGIBILITY:
Inclusion Criteria:

residual stones. recurrent stones, failed ERCP due to imacted large stone, Multiple CBD calculi with distal narrowing (Funnel syndrome), Papillary stenosis; impacted calculi, Biliary sludge-symptomatic, Sphincter of Oddi dysfunction/stenosis, Primary CBD stones; previous choledochotomy and Marked CBD dilatation.

Exclusion Criteria:

surgically unfit patients, malignancy, infections e.g, cholangitis and coagulation disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-10 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
primary outcome measure | one year
  Abd pain according to pain score from 1 to 10. total billirubin more than 1.2 mg/dl. Fever (temperature more than 38° c)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park CY, Choi SH, Kwon CI, Cho JH, Jang SI, Lee TH, Han JH, Jeong S, Ko KH. What is the better surgical treatment option for recurrent common bile duct stones? Ann Surg Treat Res. 2020 Dec;99(6):329-336. doi: 10.4174/astr.2020.99.6.329. Epub 2020 Nov 26. PMID 33304860
- [Background] Xia H, Zhang H, Xin X, Liang B, Yang T, Liu Y, Wang J, Meng X. Surgical Management of Recurrence of Primary Intrahepatic Bile Duct Stones. Can J Gastroenterol Hepatol. 2023 Jan 23;2023:5158580. doi: 10.1155/2023/5158580. eCollection 2023. PMID 36726399
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7704274/